CLINICAL TRIAL: NCT02108002
Title: Pilot Study of the Effect of Vorinostat on Nervous System Hemangioblastomas In Von Hippel-Lindau Disease
Brief Title: Effect of Vorinostat on Nervous System Hemangioblastomas in Von Hippel-Lindau Disease (Missense Mutation Only)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140067; 14-N-0067
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09-12

CONDITIONS: Von Hippel-Lindau Disease
Keywords: Missense Mutations; Hemangioblastoma; Histone Deacytelase Inhibitors; Von Hippel-Lindau Disease
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma | interventions — Vorinostat

INTERVENTIONS:
Drug: Vorinostat

SUMMARY:
Background:

- Von Hippel-Lindau (VHL) disease is a rare gene disease. People with VHL often have a brain tumor called hemangioblastoma. Standard treatment for these tumors is risky surgery. Researchers want to find new ways to treat people who have the tumors. They want to see if a drug that fights other cancers might slow the growth of hemangioblastomas in some people with VHL. Some people with VHL have mutations that make abnormal proteins. Tumors form in such people because the abnormal protein is broken down quickly. The cancer drug may work in these tumors by preventing breakdown of protein.

Objective:

- To study how the drug vorinostat affects hemangioblastomas in people with VHL.

Eligibility:

- Adults at least 18 old with hemangioblastomas from VHL.

Design:

* Participants must already be in study 03-N-0164. They must have tumor surgery scheduled.
* Participants must stop taking most medications 14 days before surgery.
* One week before surgery, participants will enter the hospital. They will be screened with medical history and physical and neurological exams. They will give blood and urine samples. Participants will have an electrocardiogram. For this test, small sticky patches are put on the arms, legs, and chest. Participants will lie still for a few minutes while a machine records heart rate and rhythm.
* Participants will take one vorinostat by mouth each day for 7 days.
* Participants will have blood drawn during the week to check for any side effects.
* Participants will have their tumor removed in surgery. Researchers will study the tumor tissue for the effects of the study drug.
* A nurse will call participants 1 month after surgery to check for side effects.

DETAILED DESCRIPTION:
Background

Central Nervous System (CNS) hemangioblastomas are the most common tumor found in the familial neoplasia syndrome, Von Hippel-Lindau (VHL).

Hemangioblastomas cause significant morbidity and mortality. While surgical resection is the treatment of choice for CNS hemangioblastomas, it is associated with morbidity and death. There is a critical need for new non-invasive treatments of VHL-associated CNS hemangioblastomas.

Vorinostat is a histone deacetylase inhibitor (HDACi) that is FDA-approved for the treatment of refractory cutaneous T-cell lymphoma (CTCL). Vorinostat has been tested in other hematologic malignancies and solid tumors. Recent data suggests that vorinostat may have a potent therapeutic effect in the treatment of VHL-associated hemangioblastomas in patients with missense germline mutations of the VHL gene. In most VHL mutation types, the abnormal VHL protein content is not active, which leads to tumor formation and growth. In missense mutation VHL disease, tumor cells contain a malformed VHL protein that is partially active. However, the protein is degraded quickly by normal cellular mechanisms. Vorinostat prevents degradation of a malformed protein within the tumors. Increased protein leads to slower growth in these tumors.

Objective

To determine whether vorinostat reduces degradation of mutant VHL protein in VHL patients with germline missense mutations.

Eligibility

Adult patients (age greater than or equal to 18 years) with a known germline missense VHL gene mutation that require surgical resection of a hemangioblastoma.

Design

We intend to conduct a pilot study with vorinostat in six patients with hemangioblastomas causing significant symptoms from tumor growth. Vorinostat will be administered if the patients are deemed surgical candidates. Patients will receive one (1) dose of 400 mg of vorinostat daily for seven (7) days prior to surgery. On the day of surgery, the patients will not receive vorinostat. Patients will undergo surgery as usual, with no change in planning or technique of the procedure. The tumor specimens from surgery will be examined for presence and quantity of mutant VHL protein. Comparisons for levels of mutant VHL protein will be made with tissue banked from previous surgical resections under 03-N-0164. Measurements of genetic expression of vascular endothelial growth factor (VEGF) and erythropoietin (EPO) will also be performed on these specimens.

Outcome Measures

1. The presence and quantity of mutant VHL protein in resected hemangioblastoma specimens, including comparison of specimens without vorinostat treatment and those with presurgical vorinostat treatment.
2. Measurement of VEGF and EPO results from resected hemangioblastoma specimens, including comparison of specimens without vorinostat treatment and those with presurgical vorinostat treatment.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Adult patients (age greater than or equal to 18 years)
  2. Known VHL disease arising from a missense mutation.
  3. Demonstrated clinical progression of CNS hemangioblastoma.
  4. Enrolled in 03-N-0164, Evaluation of Neurosurgical Disorders.
  5. Able to provide written informed consent.

EXCLUSION CRITERIA

1. Patients who have been previously treated with vorinostat.
2. Significant medical illnesses that in the investigator s opinion cannot be adequately controlled with appropriate therapy or would compromise the patient s ability to tolerate this therapy.
3. History of a second cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
4. Active infection or serious concurrent medical illness.
5. Pregnancy and breast-feeding.
6. Presence of any disease that will obscure toxicity or dangerously alter drug metabolism (such as uncontrolled diabetes, liver disease, bleeding disorder)
7. Currently receiving other investigational agents.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat, such as valproate.
9. Currently taking another HDACi, such as valproate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04-05; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
The presence and quantity of mutant VHL protein in resected hemangioblastoma specimens, including comparison of specimens without vorinostat treatment and those with presurgical vorinostat treatment. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harries RW. A rational approach to radiological screening in von Hippel-Lindau disease. J Med Screen. 1994 Apr;1(2):88-95. doi: 10.1177/096914139400100205. PMID 8790493
- [Background] Friedrich CA. Von Hippel-Lindau syndrome. A pleomorphic condition. Cancer. 1999 Dec 1;86(11 Suppl):2478-82. PMID 10630173
- [Background] Maher ER, Willatt L, Cuthbert G, Chapman C, Hodgson SV. Three cases of 16q duplication. J Med Genet. 1991 Nov;28(11):801-2. doi: 10.1136/jmg.28.11.801. No abstract available. PMID 1820771
- [Derived] Chittiboina P, Mandal D, Bugarini A, Asuzu DT, Mullaney D, Mastorakos P, Stoica S, Alvarez R, Scott G, Maric D, Elkahloun A, Zhuang Z, Chew EY, Yang C, Linehan M, Lonser RR. Proteostasis Modulation in Germline Missense von Hippel Lindau Disease. Clin Cancer Res. 2023 Jun 13;29(12):2199-2209. doi: 10.1158/1078-0432.CCR-22-3651. PMID 37018064